CLINICAL TRIAL: NCT05830968
Title: Clinical Evaluation of Safety and Efficacy of the InMode RF Pro System With the Morpheus8 Applicator for the Treatment of Mild to Severe Inflammatory Acne Vulgaris
Brief Title: Safety and Efficacy of Radio Frequency for the Treatment of Mild to Severe Inflammatory Acne
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO611175A
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Study Design Prospective, multicenter clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device treatment (Experimental): Treatment area will include affected areas over the entire face (presence of comedones, pustules, papules, nodules and cysts
  Interventions: Device: Morpheus8 Applicator Radiofrequency device

INTERVENTIONS:
Device: Morpheus8 Applicator Radiofrequency device — Eligible subjects will receive 2 treatments with the Morpheus8 according to the study protocol. All participants will return for 2 follow up visits: 4 weeks (1M FU) and 12 weeks (3M FU) after the 2nd treatment. Total expected study duration is ~6 months, depending on subject recruitment rate.

SUMMARY:
The aim of this trial is to evaluate the safety and efficacy of the InMode RF Pro System with the Morpheus8 face tip (24 pins) applicator for the treatment of mild, moderate and severe, facial acne vulgaris

DETAILED DESCRIPTION:
The aim of this trial is to evaluate the safety and efficacy of the InMode RF Pro System with the Morpheus8 face tip (24 pins) applicator for the treatment of mild, moderate and severe, facial acne vulgaris. Prospective, multicenter clinical study

ELIGIBILITY:
Inclusion Criteria:

* Subject is >16 years of age
* General good health confirmed by medical history and examination of the treated area.
* Subjects with mild to severe Acne Vulgaris, defined as a baseline IGA (Investigator's Global Assessment) score of 2, 3 or 4 and 10-100 inflammatory lesions (papules or pustules).
* The patients should be willing to comply with the study procedure and schedule, including the follow up visits, and will refrain from using any other acne treatment methods during the entire study period.
* Willing to avoid sun/UV exposure for duration of the study unless using sunscreen.
* Willing to refrain from starting or changing hormonal contraception for duration of study.
* Subject understands and is willing to sign the informed consent to participate in the study. Parental (or other) guardians must provide consent for minors under the age of 18.

Exclusion Criteria:- Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.

* Patients who are under pharmacological anti-acne therapy (isotretinoin or antibiotics) for the last 6 months.
* Use of botulinum toxin within prior 1 month.
* Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance
* Current or history of cancer, or premalignant condition in the treatment area.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Subject who are pregnant or nursing.
* Started or changed hormonal contraceptive within prior month of study.
* Subject is unwilling or unlikely to refrain from high UV exposure to face.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days.
* Any surgery in treated area within 3 months prior to treatment.
* Subject received other treatments such as light, CO2 laser or RF in the treatment area within 6 months of study start date.
* Simultaneous participation in another investigator drug or device study or completion of the follow-up phase for the primary endpoint of any previous study less than 30 days prior to the first evaluation in this study.
* Subject that has any condition that, at the investigator's discretion, renders the subject unsuitable for participation in this clinical research study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Percent of responder | Month 3
  Percent of responders, where responders are defined as subjects with at least a 50% reduction in number of inflammatory acne lesions from baseline to 12 weeks after the last treatment, as assessed by 3 independent reviewers using clinical photographs.
  Success Criteria: Success will be achieved if at least 50% of enrolled subjects are responders.

SECONDARY OUTCOMES:
Absolute change in number of inflammatory acne lesions | Month 3
  Absolute change in number of inflammatory acne lesions from baseline to 12 weeks after the last treatment, as assessed by 3 independent reviewers using clinical photographs
Percentage of subjects with a ≥2 point score improvement on the Investigators Global Assessment (IGA) scale | Month 3
  Percentage of subjects with a ≥2 point score improvement on the Investigators Global Assessment (IGA) scale at 12 weeks after the last treatment compared to baseline as assessed by three independent reviewers using clinical photographs.
Absolute change in non-inflammatory acne lesions | Month 3
  Absolute change In non-inflammatory acne lesions from baseline to 12 weeks after the last treatment, as assessed by 3 independent reviewers from clinical photographs
The rate of patient satisfaction with treatment, | Month 3
  The rate of patient satisfaction with treatment, using a 5-point Likert scale at 12 weeks after the last treatment
percent change in non-inflammatory acne lesions | Month 3
  percent change in number of inflammatory acne lesions from baseline to 12 weeks after the last treatment, as assessed by 3 independent reviewers using clinical photographs
Percent change in non-inflammatory acne lesions | Month 3
  Percent change in non-inflammatory acne lesions from baseline to 12 weeks after the last treatment, as assessed by 3 independent reviewers from clinical photographs

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Chapas, MD, Principal Investigator; Jole L Cohen, MD, Principal Investigator — Unafilliated
Locations (4):
- United States (4):
  - Avant Dermatology Aesthetics, Oro Valley, Arizona
  - AboutSkin Research, LLC, Greenwood Village, Colorado
  - UnionDerm, New York, New York
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No